CLINICAL TRIAL: NCT02759848
Title: The Role of Tuberculosis in Chronic Obstructive Lung Disease
Acronym: TROTIC
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Halil İbrahim Yakar, Halil İbrahim Yakar, Istanbul Medeniyet University
Other Study IDs: TROTIC-1234-TROTIC
Record Dates: First submitted 2016-05-01; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: The Role of Tuberculosis in COPD
Keywords: COPD, tuberculosis, mortality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- with history of TB
- without history of TB

SUMMARY:
Influence of tuberculosis (TB) on natural course of chronic obstructive lung disease (COPD) has not been well known. This study was designed to investigate the effects of history of TB on the long-term course of COPD.

DETAILED DESCRIPTION:
Patients hospitalized with COPD exacerbation were consecutively included (n=598). Cases were classified into two categories: those with a history of TB and those without. Clinical, demographic, and radiological features were meticulously recorded and patients were followed up for mortality. 93 patients (15%) had past TB. On average, patients with a history of TB were four-year younger (p=0.002). Our study revealed that patients with TB history were diagnosed with COPD five-year earlier and died five-year earlier as compared to the patients without TB. In addition, in the TB history positive group, the rate of hospital admissions per year was higher compared to the group that lacked TB history (2.46±0.26 vs. 1.56±0.88; p=0.001). The patients with TB history had higher PaCO2 and lower FEV1 (p=0.008 and p=0.069 respectively). Median survival was 24 months for patients with past TB, and was 36 months for those without. Kaplan-Meier analysis revealed that although 3-year survival rate was lower in patients with TB history, it was not statistically significant (p=0.08). Cox regression analysis showed that while factors such as age, PaCO2, hematocrit, BMI and the Charlson index affected mortality rates in COPD patients (p<0.05), prior history of TB did not seem to have a significant impact on the mortality.

Our results showed that past TB caused more hospitalizations, lower respiratory functions and higher arterial carbon dioxide levels. It was found that, though the mortality rates were similar, COPD patients with past TB was diagnosed and died five-year earlier. We conclude that history of TB has an important role in natural course of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with COPD exacerbations

Exclusion Criteria:

* Not diagnosed with COPD exacerbations

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with COPD exacerbation (tertiary care clinic)
Sampling Method: Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
all cause mortality | three years

CONTACTS AND LOCATIONS:
Overall Officials: Halil I Yakar, Md, Principal Investigator — Halil Ibrahim Yakar

IPD SHARING:
Plan to Share IPD: Undecided